CLINICAL TRIAL: NCT01474486
Title: Feasibility and Effectiveness of a Multi-Micronutrient Intervention as a Palliative Care Therapy in Patients With Congestive Heart Failure(CHF)
Brief Title: Feasibility and Effectiveness of Micronutrients as Palliative Care Therapy in Patients With Congestive Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Phoenix VA Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Diane Parrington, Deputy Associate Chief of Staff for Research, Phoenix VA Health Care System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Parrington 005
Record Dates: First submitted 2011-01-28; First posted 2011-11-18 (Estimated); Results first posted 2021-05-27 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-05

CONDITIONS: Congestive Heart Failure; Ischemic Cardiomyopathy
Keywords: thiamin; pyridoxine; vitamin D; zinc; congestive heart failure (CHF); ischemic cardiomyopathy; nutritional injury; quality of life
MeSH Terms: conditions — Heart Failure | interventions — Micronutrients; Ergocalciferols; Thiamine

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Micronutrients (Experimental): Thiamin one tablet daily provides 50 milligrams(mg) of thiamin, Vitamin B-50 one tablet daily: provides an additional 50 mg of thiamin, riboflavin, niacin, pantothenic acid and pyridoxine, 100 microgram(mcg folic acid, and 50 mcg cyanocobalamin (B12) and biotin; Vitamin D one 50,000 International Units(IU) tablet of ergocalciferol per week for two months followed by one tablet every other week for four months, and Zinc Sulfate (Zn SO4) one tablet daily at bedtime which provides 50 mg elemental zinc (220 mg Zn SO4)
  Interventions: Drug: Micronutrients

INTERVENTIONS:
Drug: Micronutrients — Thiamin one tablet daily provides 50 milligrams(mg) of thiamin, Vitamin B-50 one tablet daily: provides an additional 50 mg of thiamin, riboflavin, niacin, pantothenic acid and pyridoxine, 100 microgram(mcg folic acid, and 50 mcg cyanocobalamin (B12) and biotin; Vitamin D one 50,000 International Units(IU) tablet of ergocalciferol per week for two months followed by one tablet every other week for four months, and Zinc Sulfate (Zn SO4) one tablet daily at bedtime which provides 50 mg elemental zinc (220 mg Zn SO4)
  Other Names: ZnSO4, Vitamin B50, Ergocalciferol, & Thiamin Hydrochloride

SUMMARY:
The purpose of this project is to conduct a preliminary test of the feasibility of a multi-micronutrient intervention to improve micronutrient status, cardiac function and quality of life in Veterans with Congestive Heart Failure (CHF).

DETAILED DESCRIPTION:
Veterans with stable CHF resulting from ischemic cardiomyopathy with systolic dysfunction and an ejection fraction ≤45% and who fit the criteria of stage B, C and D 2 heart failure will be recruited. This is a one group study with Veterans serving as their own control. They will receive 50 mg thiamin, vitamin B50 and 220 mg Zn as Zn sulfate daily for 6 months. Additionally, they will receive 50,000 IU Vitamin D as ergocalciferol each week for 8 weeks then every other week for 16 weeks. Pre (baseline) and post (6 months) cardiac function will be tested with echocardiogram and cardiac MR (when applicable), biochemical measures of thiamine, pyridoxine, zinc and Vitamin D will be measured at baseline, 3 months, 6 months and one year. Quality of life will be measured using the Minnesota Living with Heart Failure questionnaire baseline, month 3,6,and one year. Nutritional assessment including a nutrition focused physical examination and three days food records will also be measured at baseline, month 3, 6 and one year.

ELIGIBILITY:
Inclusion Criteria:

* stable CHF (three months without an exacerbation or major change in medication regimen and cardiology provider determined medication regimen (angiotensin II receptor blockers (ARBs), aldosterone, angiotensin converting enzyme (ACE) inhibitors and Beta blockers) has been maximized), Stage B, C or D CHF resulting from ischemic cardiomyopathy with an ejection fraction ≤ 45% with or without a pacemaker or defibrillator . Potential participants who require further medication titration to attain maximal benefit, will need to wait 30 days after the provider has maximized the dose of medication to participate.

Exclusion Criteria:

* recent (within the last three months) acute myocardial infarction, or unstable angina, pacemaker or defibrillator placed less than six months prior, or anticipated pacemaker or defibrillator placement in the next six months, or a bi ventricular pacemaker, corticosteroid use (> 20 mg Prednisone use or its equivalent per day > 2 weeks duration), isoniazid therapy, use of the study nutrition supplements at the study doses for the past month or longer,(if the participant has been taking a multivitamin or multivitamin with minerals , or other water soluble vitamins they will need to stop taking these for at least one month prior to initiating the study intervention), end-stage liver disease, end-stage renal disease requiring dialysis, receiving chemotherapy or radiation therapy, active alcohol/ substance abuse, pregnancy /lactation, women of childbearing potential who do not have medical documentation of surgically induced menopause, pancreatitis, any psychological issues like severe depression, claustrophobia, active problematic post-traumatic stress disorder (PTSD), or memory loss that prevents compliance with the supplement intake, agoraphobia which may interfere attendance at research visits or fear of needles which would limit their ability to have the blood tests completed, and any active eating disorders. Cardiac Magnetic Resonance Imaging (MRI) scan will not be used to test cardiac function in participants with a pacemaker or defibrillator. Nor will it be used for potential subjects with ferro magnetic materials (i.e., penile stimulator), inability to lie flat for up to one hour, inability to hold their breath for up to 15 seconds or those with claustrophobia.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-04; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diane J Parrington, PhD, Principal Investigator — Phoenix VA Health Care System
Locations (1):
- Phoenix VA Health Care System, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 40 participants consented to the study. Twelve were screen failures and six withdrew following consent but prior to their first visit when baseline data collection would have taken place and the intervention would have started. Therefore twenty-two participants received the intervention.
  The participants served as their own control, so there is only one arm of the study.
Period: Overall Study
Arm/Group | Micronutrients
Started | 28
Treated | 22
Completed | 20
Not Completed | 8
Not completed — Death | 2
Not completed — Withdrawal by Subject | 4
Not completed — Withdrawn by the PI: One didn't understand what he consented for and one required surgery. | 2

BASELINE CHARACTERISTICS:
Arm/Group | Micronutrients
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 10
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 64.0 [59.0 to 75.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 22
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 2
  Caucasian | 19
  Hispanic | 1
Region of Enrollment [Number; unit: participants]
  United States | 22
Minnesota Living with Heart Failure Questionnaire [Median (Inter-Quartile Range); unit: units on a scale] — Total score on the Minnesota Living with Heart Failure Questionnaire. The scale is used to determine how much heart failure has affected life during the past month. There are 21 questions, each with 5 possible answers 0-5 where 0 is No or not applicable, and 1 is Very Little and 5 is Very Much. The lowest possible score is 0 and the highest possible score is 105. A low score indicates heart failure has little affect on quality of life and a high score indicates heart failure is negatively affecting quality of life.
  Participants completed the questionnaire during the research visits.
  units on a scale | 15.0 [4.0 to 48.0]
Serum vitamin B1 [Median (Inter-Quartile Range); unit: nmoL/L] — Serum B1 or thiamin was measured in nmoL/L. The reference range was 78-185 nmoL/L.
  nmoL/L | 122 [114 to 134]
Serum B6 [Median (Inter-Quartile Range); unit: ng/mL] | 7.6 [5.0 to 10.4]
Serum Zinc [Median (Inter-Quartile Range); unit: mcg/dL] | 76.0 [63.0 to 87.0]
Serum Vitamin D [Median (Inter-Quartile Range); unit: ng/mL] | 32.1 [24.6 to 37.0]

OUTCOME MEASURES:

1. Primary Outcome: Change in Left Ventricular Ejection Fraction by Echocardiogram
Description: Change in Left Ventricular Ejection Fraction (LVEF) by Echocardiogram. The measure is the difference between the LVEF at 6 months from the baseline LVEF. A higher LVEF shows improvement and a lower LVEF shows worsening.
Time Frame: Change from baseline in Left Ventricular Ejection Fraction at 6 months
Population: All individuals in whom either baseline or 6 month measures were obtained.
Measure: Least Squares Mean (Standard Error); unit: Percent
Groups:
- Micronutrients: Thiamin one tablet daily provides 50 milligrams(mg) of thiamin, Vitamin B-50 one tablet daily: provides an additional 50 mg of thiamin, riboflavin, niacin, pantothenic acid and pyridoxine, 100 microgram(mcg folic acid, and 50 mcg cyanocobalamin (B12) and biotin; Vitamin D one 50,000 International Units(IU) tablet of ergocalciferol per week for two months followed by one tablet every other week for four months, Zinc Sulfate (Zn SO4) one tablet daily at bedtime which provides 50 mg elemental zinc (220 mg Zn SO4)
  Micronutrients: Thiamin one tablet daily provides 50 milligrams(mg) of thiamin, Vitamin B-50 one tablet daily: provides an additional 50 mg of thiamin, riboflavin, niacin, pantothenic acid and pyridoxine, 100 microgram(mcg folic acid, and 50 mcg cyanocobalamin (B12) and biotin; Vitamin D one 50,000 International Units(IU) tablet of ergocalciferol per week for two months followed by one tablet every other week for four months, and Zinc Sulfate (Zn SO4) one tablet daily at b
Arm/Group | Micronutrients
Number analyzed (Participants) | 21
Percent | 1.1 (2.3)
Statistical Analysis 1: Comparison: Micronutrients; Test type: Other; p = 0.64, Mixed Models Analysis

2. Primary Outcome: Change in Left Ventricular Ejection Fraction as Measured by Magnetic Resonance Imaging (MRI)
Description: Left Ventricular Ejection Fraction Measured by Magnetic Resonance Imaging (MRI). The measure is the difference between the LVEF at 6 months from the baseline LVEF. A higher LVEF shows improvement and a lower LVEF shows worsening.
Time Frame: Change from baseline in Left Ventricular Ejection Fraction at 6 months
Population: All persons with at least one measurement of LVEF by MRI.
Measure: Least Squares Mean (Standard Error); unit: Percent
Groups:
- Micronutrients: Micronutrients: Thiamin 1 tablet daily provides 50 milligrams(mg) of thiamin, Vitamin B-50 1 tablet daily: provides 50 mg of thiamin, riboflavin, niacin, pantothenic acid & pyridoxine, 100 microgram (mcg) folic acid, & 50 mcg cyanocobalamin (B12) & biotin; Vitamin D 1 50,000 International Units(IU) tablet of ergocalciferol per week for 2 months followed by 1 tablet every other week for 4 months, and Zinc Sulfate (Zn SO4) 1 tablet daily at bedtime which provides 50 mg elemental zinc (220 mg Zn SO4)
Arm/Group | Micronutrients
Number analyzed (Participants) | 13
Percent | 3.8 (3.4)

3. Secondary Outcome: Change in Quality of Life
Description: The "Minnesota Living with Heart Failure Questionnaire" was used to assess quality of life (QOL). This scale has 21 questions and each question has a possible score of 0 -5, where 0 is no or not applicable, 1 is very little and 5 is very much. The score for each question measures how much heart failure is affecting QOL. The higher the score the more heart failure is affecting QOL. Possible range of total scores is 0 - 105. The change from baseline QOL to quality of life at 3 months was calculated by subtracting the 3 month score from the baseline score. A lower score at 3 months indicates better QOL and a high score at 3 months indicates a worse QOL.
Time Frame: Change from baseline Quality of Life at 3 months
Population: All individuals with either baseline or 3 month measure of Quality of Life.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Micronutrients: Thiamin one tablet daily provides 50 milligrams(mg) of thiamin, Vitamin B-50 one tab daily: provides an additional 50 mg of thiamin, riboflavin, niacin, pantothenic acid and pyridoxine, 100 microgram(mcg folic acid, and 50 mcg cyanocobalamin (B12) and biotin; Vitamin D one 50,000 International Units(IU) tab of ergocalciferol per week for two months followed by one tab every other week for four months, and Zinc Sulfate (Zn SO4) one tabdaily at bedtime which provides 50 mg elemental zinc (220 mg Zn SO4)
  Micronutrients: Thiamin one tab daily provides 50 milligrams(mg) of thiamin, Vitamin B-50 one tab daily: provides an additional 50 mg of thiamin, riboflavin, niacin, pantothenic acid and pyridoxine, 100 microgram(mcg folic acid, and 50 mcg cyanocobalamin (B12) and biotin; Vitamin D one 50,000 International Units(IU) tab of ergocalciferol per week for two months followed by one tab every other week for four months, and Zinc Sulfate (Zn SO4) one tablet daily at bedtime which provides 50
Arm/Group | Micronutrients
Number analyzed (Participants) | 22
units on a scale | -8.3 (6.9)

4. Secondary Outcome: Nutritional Status
Description: Nutritional Injury (NI) stage was used to assign nutritional status. Nutritional injury describes the interaction between agent, host and environmental factors as 6 progressive stages of altered nutritional status leading to nutritional disease. The 6 stages are seen as progressive beginning with (1) adaptation and diminishing or exceeding reserves, (2) reserves exhausted/ exceeded, (3) physiologic and metabolic alterations related to under/over nutrition, (4) non-specific signs and symptoms of under/over nutrition, (5) illness / specific signs and symptoms of under/over nutrition and (6) permanent damage/damage unresponsive to treatment. The following were used to determine overall nutritional status: body mass index, diet quality, blood nutrient levels and other biochemical measures, physical signs and symptoms of nutrient deficiencies or excesses. The lower the stage the less nutritional injury. The outcome measure is the difference in NI from baseline at 3 months.
Time Frame: Change from baseline in nutritional status at 3 months
Population: All with both baseline and 3 month assessment of nutritional status
Measure: Median (Inter-Quartile Range); unit: score on a scale
Groups:
- Micronutrients: Thiamin one tablet daily provides 50 milligrams(mg) of thiamin, Vitamin B-50 one tab daily: provides an additional 50 mg of thiamin, riboflavin, niacin, pantothenic acid and pyridoxine, 100 microgram(mcg) folic acid, and 50 mcg cyanocobalamin (B12) and biotin; Vitamin D one 50,000 International Units(IU) tab of ergocalciferol per week for two months followed by one tab every other week for four months, and Zinc Sulfate (Zn SO4) one tab daily at bedtime which provides 50 mg elemental zinc (220 mg Zn SO4)
  Micronutrients: Thiamin one tab daily provides 50 mg of thiamin, Vitamin B-50 one tab daily: provides an additional 50 mg of thiamin, riboflavin, niacin, pantothenic acid and pyridoxine, 100 mcg folic acid, and 50 mcg cyanocobalamin (B12) and biotin; Vitamin D one 50,000 IU tab of ergocalciferol per week for two months followed by one tab every other week for four months, and Zinc Sulfate (Zn SO4) one tab daily at bedtime which provides 50 mg elemental zinc (220 mg Zn SO4)
Arm/Group | Micronutrients
Number analyzed (Participants) | 22
score on a scale | 0 [-1 to 0]

5. Secondary Outcome: Change in Quality of Life
Description: The "Minnesota Living with Heart Failure Questionnaire" was used to assess quality of life (QOL). This scale has 21 questions and each question has a possible score of 0 - 5, where 0 is no or not applicable, 1 is very little and 5 is very much. The score for each question measures how much heart failure is affecting QOL. The higher the score the more heart failure is affecting QOL. Possible range of total scores is 0 - 105. The change from baseline QOL to quality of life at 6 months was calculated by subtracting the 6 month score from the baseline score. A lower score at 6 months indicates better QOL and a higher score at 6 months indicates a worse QOL.
Time Frame: Change from baseline quality of life at 6 months
Population: All individuals with either a baseline or six month measure of Quality of Life.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Micronutrients
Number analyzed (Participants) | 22
units on a scale | -5.9 (7.0)

6. Secondary Outcome: Change on Quality of Life
Description: The "Minnesota Living with Heart Failure Questionnaire" was used to assess quality of life (QOL). This scale has 21 questions and each question has a possible score of 0 - 5, where 0 is no or not applicable, 1 is very little and 5 is very much. The score for each question measures how much heart failure is affecting QOL. The higher the score the more heart failure is affecting QOL. Possible range of total scores is 0 - 105. The change from baseline QOL to quality of life at 12 months was calculated by subtracting the 12 month score from the baseline score. A lower score at 12 months indicates better QOL and a higher score at 12 months indicates a worse QOL.
Time Frame: Change from baseline quality of life at 12 months
Population: All in whom either Baseline or 12 month Quality of Life was assessed.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Micronutrients
Number analyzed (Participants) | 22
units on a scale | 2.6 (8.8)

7. Secondary Outcome: Nutritional Status
Description: Nutritional Injury (NI) stage was used to assign nutritional status. Nutritional injury describes the interaction between agent, host and environmental factors as 6 progressive stages of altered nutritional status leading to nutritional disease. The 6 stages are seen as progressive beginning with (1) adaptation and diminishing or exceeding reserves, (2) reserves exhausted/ exceeded, (3) physiologic and metabolic alterations related to under/over nutrition, (4) non-specific signs and symptoms of under/over nutrition, (5) illness / specific signs and symptoms of under/over nutrition and (6) permanent damage/damage unresponsive to treatment. The following were used to determine overall nutritional status: body mass index, diet quality, blood nutrient levels and other biochemical measures, physical signs and symptoms of nutrient deficiencies or excesses. The lower the stage the less nutritional injury. The outcome measure is the difference in NI from baseline at 6 months.
Time Frame: Change from baseline in nutritional status at 6 months
Population: All individuals with both baseline and 6 month assessment of nutritional status.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Groups:
- Micronutrients: Thiamin one tablet daily provides 50 milligrams(mg) of thiamin, Vitamin B-50 one tab daily: provides an additional 50 mg of thiamin, riboflavin, niacin, pantothenic acid and pyridoxine, 100 microgram(mcg) folic acid, and 50 mcg cyanocobalamin (B12) and biotin; Vitamin D one 50,000 International Units(IU) tab of ergocalciferol per week for two months followed by one tab every other week for four months, and Zinc Sulfate (Zn SO4) one tab daily at bedtime which provides 50 mg elemental zinc (220 mg Zn SO4)
  Micronutrients: Thiamin one tab daily provides 50 mg of thiamin, Vitamin B-50 one tab daily: provides an additional 50 mg of thiamin, riboflavin, niacin, pantothenic acid and pyridoxine, 100 mcg folic acid, and 50 mcg cyanocobalamin (B12) and biotin; Vitamin D one 50,000 IU tablet of ergocalciferol per week for two months followed by one tablet every other week for four months, and Zinc Sulfate (Zn SO4) one tablet daily at bedtime which provides 50 mg elemental zinc (220 mg Zn SO4)
Arm/Group | Micronutrients
Number analyzed (Participants) | 20
score on a scale | 0 [-0.5 to 0]

8. Secondary Outcome: Nutritional Status
Description: Nutritional Injury (NI) stage was used to assign nutritional status. Nutritional injury describes the interaction between agent, host and environmental factors as 6 progressive stages of altered nutritional status leading to nutritional disease. The 6 stages are seen as progressive beginning with (1) adaptation and diminishing or exceeding reserves, (2) reserves exhausted/ exceeded, (3) physiologic and metabolic alterations related to under/over nutrition, (4) non-specific signs and symptoms of under/over nutrition, (5) illness / specific signs and symptoms of under/over nutrition and (6) permanent damage/damage unresponsive to treatment. The following were used to determine overall nutritional status: body mass index, diet quality, blood nutrient levels and other biochemical measures, physical signs and symptoms of nutrient deficiencies or excesses. The lower the stage the less nutritional injury. The outcome measure is the difference in NI from baseline at 12 months.
Time Frame: Change from baseline in nutritional status at 12 months
Population: All individuals with both baseline and 12 month assessments of nutritional status.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Micronutrients
Number analyzed (Participants) | 15
score on a scale | 0 [0 to 0]

ADVERSE EVENTS:
Time Frame: The data was collected from the time of consent until the final visit, which occurred either six months or one year after starting the intervention. The protocol was amended to include data six months post-intervention, but not all participants continued on for the full year.
Description: The adverse events were collected during patient visits. In the cases with abnormal lab values, select lab results (whole blood thiamin and plasma pyridoxine) were not available for up to two weeks following the visit. When the thiamin or pyridoxine were abnormal (defined as above the reference range) they reflected compliance with the study intervention not toxicity.
Arm/Group | Micronutrients
All-Cause Mortality (participants affected / at risk) | 2/22
Serious Adverse Events (participants affected / at risk) | 8/22
Other Adverse Events (participants affected / at risk) | 16/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Micronutrients (N=22)
All Cause Mortality (Cardiac disorders) | 1 (1) — CHF exacerbation following Non-ST segment elevation myocardial infarction
All cause mortality (Cardiac disorders) | 1 (1) — Admitted into and expired at community hospital. Cause is unknown. Participant had contacted the VA within 3 days of his death complaining of excessive dizziness.
Serious Adverse Event (Cardiac disorders) | 1 (2) — Inpatient hospitalization for pain caused by ischemia of right lower extremity. Second hospitalization for bifemoral bypass of the right lower extremity.
Serious Adverse Events (Infections and infestations) | 1 (3) — One inpatient hospitalization for wound dehiscence of L anterior ankle wound 9 months s/p L total ankle replacement. Second admission one month later for cellulitis of same area, followed by a 3rd hospitalization for same diagnoses 3 months later.
Serious Adverse Event (Infections and infestations) | 1 (1) — Inpatient hospitalization for LLE cellulitis secondary to leg trauma.
Adverse Events (Gastrointestinal disorders) | 1 (1) — Inpatient hospitalization for small bowel obstruction and ileus.
Serious Adverse Event (Infections and infestations) | 1 (1) — Hospitalization for bacteremia from a urinary source. Also had an obstructing urethral stone.
Serious Adverse Event (General disorders) | 1 (1) — Admitted for dehydration due to medication overuse.
Serious Adverse Event (Blood and lymphatic system disorders) | 1 (1) — Hospital admission for uncontrolled bleeding and anemia after lacerating his arm. This is the same participant as described in #5.
Serious Adverse Event (Vascular disorders) | 1 (1) — Hospitalized for a Left Lower Extremity femoral bypass graft thrombosis. This occurred between consent and starting the intervention and is the same participant at #2.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Micronutrients (N=22)
Other (Metabolism and nutrition disorders) | 12 (17) — Abnormal lab value
Other (Gastrointestinal disorders) | 2 (2) — Diarrhea
Other (Eye disorders) | 2 (2) — Conjunctivitis
Other (General disorders) | 2 (2) — Flu-like symptoms

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes